CLINICAL TRIAL: NCT04003597
Title: 'Low-salt' Bread as Part of a Pragmatic Reduced-salt Diet for Lowering Blood Pressure in Adults With Elevated Blood Pressure
Brief Title: 'Low-salt' Bread as a Means of Reducing Dietary Salt and Lowering Blood Pressure
Acronym: Saltbreads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Kevin D. Cashman, Professor of Food and Health, University College Cork
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 06/rd/c/455
Record Dates: First submitted 2019-06-21; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Elevated Blood Pressure
Keywords: Low-salt bread; Dietary sodium restriction; Pre-hypertension; Hypertension stage 1
MeSH Terms: conditions — Hypertension; Prehypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The biochemical outcome measures were assessed by researchers masked to the phase of the cross-over intervention from which the samples were derived.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual-salt diet (Placebo Comparator): Usual-salt diet followed for 5 weeks
  Interventions: Other: Usual-salt diet
- Reduced-salt diet (Active Comparator): Reduced-salt diet followed for 5 weeks
  Interventions: Other: Reduced-salt diet

INTERVENTIONS:
Other: Usual-salt diet — Subjects followed their usual-salt diet but were asked to consume an equivalent in-house produced brown or white sliced pan bread equivalent in composition to the low-salt version but with its more typical salt content (1.2 g/100 g).
  Arms: Usual-salt diet
Other: Reduced-salt diet — Subjects randomized to start on the reduced-salt diet were asked to restrict their consumption of dietary salt using a combination of pragmatic dietary advice as well as the replacement of bread and a limited number of other foods with equivalent foods which had lower salt content; these were provided to the participants. At the beginning of the salt restriction period, a research nutritionist provided the subjects with a list of the common salt-containing food (salted and naturally salty) and were asked to limit the consumption of such, as feasible. The subjects received in-house prepared 'low-salt (<0.3 g/100 g)' brown or white sliced pan bread as well as no-salt margarine/butter, and were given luncheon meats with no added salt if desired (optional).
  Arms: Reduced-salt diet

SUMMARY:
In the context of public health, reformulation of bread in terms of salt content remains an important measure to help achieve a reduction in salt intake in the population. Therefore, the aim of this study was to examine, using a 5-week cross-over design, food-based intervention trial, the potential for inclusion of 'low-salt' bread as part of a pragmatic reduced-salt diet on blood pressure (BP) in adults with slightly to moderately elevated BP.

The study consisted of a randomized crossover trial of the effect of reduced-salt intake or usual-salt intake for 5 weeks on BP (as the primary outcome) in adults with slightly to moderately elevated BP (seated office systolic BP >120 and <160 mmHg or a diastolic BP >80 and <95 mmHg; identified by a pre-screening phase).

Subjects were randomly assigned to the reduced-salt diet or their usual-salt diet (control) for 5 weeks, followed by crossover to the alternative dietary regimen for a further 5 weeks. Subjects randomized to start on the reduced-salt diet were asked to restrict their consumption of dietary salt using a combination of pragmatic dietary advice as well as the replacement of bread and a limited number of other foods with equivalent foods which had lower salt content; these were provided to the participants. At the beginning of the salt restriction period, a research nutritionist provided the subjects with a list of the common salt-containing food and were asked to limit the consumption of such, as feasible. The subjects received in-house prepared 'low-salt (<0.3 g/100 g)' brown or white sliced pan bread as well as no-salt margarine/butter, and were given luncheon meats with no added salt, if desired (optional); these were supplied regularly by the research staff. Subjects commencing the trial on the control diet were allowed to follow their usual diet but were asked to consume an in-house produced brown or white sliced pan bread equivalent in composition to the low-salt version but with its more typical salt content (1.2 g/100 g).

Participants met the research staff weekly to receive breads and no-salt margarine/butter as well as luncheon meats (where applicable), and at these meetings the staff promoted compliance with the intervention and encouraged completion of the study protocol.

BP and other assessments were made at baseline and at the end of week 5 and week 10.

DETAILED DESCRIPTION:
Brief background and context for the study:

The World Health Organization's Global Action Plan for the Prevention and Control of Non-Communicable Disease includes a voluntary global target of a 30% relative reduction in mean population intake of salt/sodium by 2025. Bread and cured/processed meats collectively contribute anything from about a third upwards of total salt intake of adults in many Western countries. Reformulation of bread in terms of salt content remains an important measure to help achieve a reduction in salt intake in the population. Therefore, the aim of this study was to examine, using a 5-week cross-over design, food-based intervention trial, the potential for inclusion of 'low-salt' bread as part of a pragmatic reduced-salt diet on blood pressure (BP) in adults with slightly to moderately elevated BP.

Design:

The study consisted of a randomized crossover trial of the effect of reduced-salt intake or usual-salt intake for 5 weeks on BP (primary outcome) and biochemical markers of calcium and bone metabolism as well as plasma lipids (secondary outcomes) in adults with slightly to moderately elevated BP.

Potential volunteers were screened for BP over 3 weeks preceding the intervention phase of the trial during which seated office systolic and diastolic BP were measured weekly and those with systolic BP >120 and <160 mmHg or a diastolic BP >80 and <95 mmHg were considered eligible.

The dietary intervention phase of the trial was designed in two successive dietary periods, each of 5 weeks. Subjects were randomly assigned to the reduced-salt diet or their usual-salt diet (control) for 5 weeks, followed by crossover to the alternative dietary regimen for a further 5 weeks. At baseline (week 0), the subjects visited the Human Nutrition Studies Unit within University College Cork in a fasting state and had their BP measured. Prior to the baseline visit, subjects received instructions on how to collect a 24-h urine sample and were provided with a suitable container for collection. On the day of the baseline visit, subjects brought the 24-h urine sample collected from the previous day and deposited it in a cold room area dedicated for such collections. A blood sample was taken from each subject between 08.30 am and 10.30 am by a trained phlebotomist and anthropometric measures including height and weight, were taken. A health and lifestyle questionnaire, which assessed physical activity, general health, smoking status and alcohol consumption was completed by each subject. Subjects randomized to start on the reduced-salt diet were asked to restrict their consumption of dietary salt using a combination of pragmatic dietary advice as well as the replacement of bread and a limited number of other foods with equivalent foods which had lower salt content; these were provided to the participants. At the beginning of the salt restriction period, a research nutritionist provided the subjects with a list of the common salt-containing food and were asked to limit the consumption of such, as feasible. The subjects received in-house prepared 'low-salt (<0.3 g/100 g)' brown or white sliced pan bread as well as no-salt margarine/butter, and were given luncheon meats with no added salt, if desired (optional). Subjects commencing the trial on the control diet were allowed to follow their usual diet but were asked to consume an in-house produced brown or white sliced pan bread equivalent in composition to the low-salt version but with its more typical salt content (1.2 g/100 g).

During the intervention phase, each participant made 2 further visits to the study unit, one each on the last day of dietary period 1 (week 5) and dietary period 2 (week 10). At these visits, BP measurements were taken as well as other anthropometric measures, including height and weight. An overnight fasting blood sample was also taken from each participant between 08.30 am and 10.30 am by a trained phlebotomist, and on each of the visits, the subjects provided a 24-hour urine sample collected the previous day. Following blood sampling the participants received their breakfast.

Participants met the research staff weekly to receive breads and no-salt margarine/butter as well as luncheon meats (where applicable), and at these meetings the staff promoted compliance with the intervention and encouraged completion of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* consenting adult Caucasian men and women, aged ≤65 y;
* a seated office systolic BP >120 and <160 mmHg and/or a diastolic BP >80 and <95 mmHg (based on the mean BP across 3 screening visits as part of a pre-intervention phase of the trial)
* willing to consume study breads

Exclusion Criteria:

* taking anti-hypertensive medication;
* taking any medications known to interfere with blood pressure or calcium or bone metabolism;
* Severe medical illness;
* celiac disease;
* hypercalcemia;
* known intestinal malabsorption syndrome,
* excessive alcohol use (>14 drinks/week);
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-01-03 (Actual); Primary Completion 2010-07-30 (Actual); Study Completion 2010-07-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure at end of intervention periods | After 5 weeks of intervention
  Measured as seated office systolic blood pressure at end of usual salt dietary period and at end of reduced-salt dietary period

SECONDARY OUTCOMES:
Diastolic blood pressure | After 5 weeks of intervention
  Measured as seated office diastolic blood pressure at end of usual salt dietary period and at end of reduced-salt dietary period
Urinary Calcium | After 5 weeks of intervention
  Assessed in 24-hour urine collected at end of usual salt dietary period and at end of reduced-salt dietary period
Urinary N-telopeptides of Type I collagen | After 5 weeks of intervention
  Biomarker of bone resorption; Assessed in 24-hour urine collected at end of usual salt dietary period and at end of reduced-salt dietary period
Serum Parathyroid Hormone | After 5 weeks of intervention
  Index of calcium metabolism; Assessed in 24-hour urine collected at end of usual salt dietary period and at end of reduced-salt dietary period
Serum C-telopeptide of Type I collagen | After 5 weeks of intervention
  Biomarker of bone resorption; Assessed in 24-hour urine collected at end of usual salt dietary period and at end of reduced-salt dietary period
Serum Osteocalcin | After 5 weeks of intervention
  Biomarker of bone formation; Assessed in fasting serum collected at end of usual salt dietary period and at end of reduced-salt dietary period
Serum Bone-specific alkaline phosphatase | After 5 weeks of intervention
  Biomarker of bone formation; Assessed in fasting serum collected at end of usual salt dietary period and at end of reduced-salt dietary period
Plasma triglycerides | After 5 weeks of intervention
  Index of circulating lipids and CHD risk; Assessed in fasting plasma collected at end of usual salt dietary period and at end of reduced-salt dietary period
Serum total-cholesterol | After 5 weeks of intervention
  Index of circulating lipids and CHD risk; Assessed in fasting plasma collected at end of usual salt dietary period and at end of reduced-salt dietary period
Plasma LDL-cholesterol, | After 5 weeks of intervention
  Index of circulating lipids and CHD risk; Assessed in fasting plasma collected at end of usual salt dietary period and at end of reduced-salt dietary period
Plasma HDL-cholesterol | After 5 weeks of intervention
  Index of circulating lipids and CHD risk; Assessed in fasting plasma collected at end of usual salt dietary period and at end of reduced-salt dietary period

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Cashman, PhD, Principal Investigator — University College Cork
Locations (1):
- School of Food and Nutritional Sciences, University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No